CLINICAL TRIAL: NCT02328170
Title: Comparative Study of Specific IgE Levels to Common Foods and Aeroallergens Among Thai Children Measured by EUROIMMUN Allergy and ImmunoCap
Brief Title: Comparative Study of Specific IgE Levels to Common Foods and Aeroallergens Measured by EUROIMMUN Allergy and ImmunoCap
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, JITTIMA VESKITKUL, Asst.Prof., Mahidol University
Other Study IDs: 054/2557(EC2)
Record Dates: First submitted 2014-12-11; First posted 2014-12-31 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Allergy
Keywords: immunoglobulin E, food hypersensitivities, child, allergens
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Clotted blood 3 mL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUROIMMUN Allergy: Immunoblot assay
  Interventions: Other: EUROIMMUN Allergy
- ImmunoCap: Fluoroallergosorbent test
  Interventions: Other: ImmunoCap

INTERVENTIONS:
Other: EUROIMMUN Allergy — Immunoblot assay
  Groups: EUROIMMUN Allergy
Other: ImmunoCap — Fluoroallergosorbent test
  Groups: ImmunoCap

SUMMARY:
The purpose of this study is to determine the correlation of specific IgE levels to common foods and aeroallergens measured by EUROIMMUN Allergy and ImmunoCap

DETAILED DESCRIPTION:
Children aged 0-15 years old who was diagnosed as asthma and/or allergic rhinitis, atopic dermatitis, food allergy, and underwent to measured specific IgE levels to suspicious relevant allergen, were invited to join the study.

Specific IgE levels of each patient was measured by EUROIMMUN Allergy and ImmunoCap.

The levels of specific IgE to Dermatophagoides pteronyssinus, Dermatophagoides farinae, American cockroach, Bermuda, Johnson, Cat dander, Cow's milk, Egg white and wheat were determined the correlation between these two methods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed as asthma and/or allergic rhinitis and/or atopic dermatitis and/or food allergy and have to measured specific IgE levels to relevant allergens

Exclusion Criteria:

* Having underlying disease including cardiovascular disease, chronic lung disease and immunodeficiency disease
* Denied to enrolled to the study

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who was diagnosed as having asthma and/or allergic rhinitis and/or atopic dermatitis and/or food allergy, were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
specific IgE levels measured by EUROIMMUN Allergy and ImmunoCap | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Jittima Veskitkul, Assist Prof., Principal Investigator — Mahidol University
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No